CLINICAL TRIAL: NCT02355093
Title: Adductor Canal Block Versus Femoral Nerve Block for Analgesia After Anterior Cruciate Ligament Reconstruction Arthroscopically
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Shanghai Jiao Tong University Affiliated Sixth People's Hospital (Other)
Responsible Party: Principal Investigator, Daqiang Zhao, Daqiang Zhao, Shanghai Jiao Tong University Affiliated Sixth People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ACB vs FNB
Record Dates: First submitted 2015-01-28; First posted 2015-02-04 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-01

CONDITIONS: Anesthesia; Reaction
MeSH Terms: interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- adductor canal block (ACB) (Experimental): We performed an ultrasound survey at the medial part of the thigh，the needle is introduced in-plane and 2 to 3 mL of saline is used to ensure correct placement of the needle in the vicinity of the saphenous nerve in the adductor canal,the catheter is introduced and advanced 1 to 2 cm beyond the tip of the needle.The study medication is administered as an infusion of 0.2% ropivacaine at a rate of 5mL/h during the next 48 hours.
  Interventions: Procedure: adductor canal block (ACB); Drug: ropivacaine
- Femoral nerve block (FNB) (Active Comparator): the catheter is inserted in-plane with the probe parallel to the inguinal crease, to obtain a short-axis view of the nerve. The correct needle placement is confirmed by injecting 2 to 3 mL of saline to cause tissue expansion below the iliac fascia, lateral to the femoral artery, and in the vicinity of the femoral nerve. The catheter is introduced 1 to 2 cm beyond the tip of the needle，an infusion of 0.2% ropivacaine at a rate of 5mL/h is administered during the next 48 hours.
  Interventions: Procedure: Femoral nerve block (FNB); Drug: ropivacaine

INTERVENTIONS:
Procedure: adductor canal block (ACB) — We performed an ultrasound survey at the medial part of the thigh，the needle is introduced in-plane and 2 to 3 mL of saline is used to ensure correct placement of the needle in the vicinity of the saphenous nerve in the adductor canal,the catheter is introduced and advanced 1 to 2 cm beyond the tip of the needle.The study medication is administered as an infusion of 0.2% ropivacaine at a rate of 5mL/h during the next 48 hours.
  Arms: adductor canal block (ACB)
Procedure: Femoral nerve block (FNB) — the catheter is inserted in-plane with the probe parallel to the inguinal crease, to obtain a short-axis view of the nerve. The correct needle placement is confirmed by injecting 2 to 3 mL of saline to cause tissue expansion below the iliac fascia, lateral to the femoral artery, and in the vicinity of the femoral nerve. The catheter is introduced 1 to 2 cm beyond the tip of the needle，an infusion of 0.2% ropivacaine at a rate of 5mL/h is administered during the next 48 hours.
  Arms: Femoral nerve block (FNB)
Drug: ropivacaine

SUMMARY:
This study aims to compare continuous femoral nerve block with adductor canal block after anterior cruciate ligament reconstruction arthroscopically，especially in the effect on quadriceps strength; and to evaluate which regional anesthesia is more ideal for the patients postoperatively.

DETAILED DESCRIPTION:
Forty patients with American Society of Anesthesiologists（ASA） Ⅰ-Ⅲ（no limitation of age and gender）are randomized to receive either a continuous adductor canal block(ACB) or a femoral nerve block(FNB) via a catheter (a continuous infusion of 0.2% ropivacaine, 5 mL/h for 48 hours)in the PACU immediately after the anterior cruciate ligament reconstruction arthroscopically. Patients were under general anesthesia during the operation and received a femoral nerve block with 0.25% ropivacaine 10ml before the surgery.Both groups will receive postoperatively IV patient controlled analgesia (PCA) with morphine (bolus 0.8mg,lock-out time 15 minutes, background infusion 2ml/h)beside the continuous nerve block. Patients are going to be visited for follow-up on the day of surgery and in the following two days. Quadriceps strength is assessed with the displacement of patella.VAS at rest time、degree of knee flexion、VAS at 45°flexion of the knee、dose of opioids、whether the patient has sleep disturbance are also recorded.

ELIGIBILITY:
Inclusion Criteria:

* ASA Ⅰ-Ⅲ
* Anterior Cruciate Ligament Reconstruction

Exclusion Criteria:

* patient refusal
* chronic use of opioids
* coagulation disorders
* infection at the puncture site
* allergic to anaesthetic
* preexisting neurological disorders
* communication difficulties

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-07; Primary Completion 2015-03 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
quadriceps muscle strength, as measured by handheld dynamometer. | 3 days

SECONDARY OUTCOMES:
pain at rest time and during flexion of the knee, as measured by visual analog score(VAS). | 3 days

OTHER OUTCOMES:
Dose of opioids | 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Daqiang Zhao, Master, Principal Investigator — Shanghai Jiaotong University Affiliated Sixth People's Hospital Shanghai,China